CLINICAL TRIAL: NCT02445729
Title: Impact of Timing of Wound Dressing Removal After Cesarean Section: Effect of Dressing Removal at 24 Hours Versus 48 Hours on Wound Healing and Incidence of Surgical Site Infections Following Cesarean Section
Brief Title: Impact of Timing of Wound Dressing Removal After Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital (Other); Dicle University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-0548
Record Dates: First submitted 2015-05-12; First posted 2015-05-15 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2019-06

CONDITIONS: Abdominal Wall Wound
Keywords: Cesarean Section; Wound Healing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dressing Removal at 24 Hours (Active Comparator): These patients are randomly assigned to have their dressing removed 24 hours after cesarean section.
  Interventions: Other: Dressing removal at 24 hours
- Dressing Removal at 48 Hours (Active Comparator): These patients are randomly assigned to have their dressing removed 48 hours after cesarean section.
  Interventions: Other: Dressing removal at 48 hours

INTERVENTIONS:
Other: Dressing removal at 24 hours — Dressing will be removed 24 hours after cesarean section and wounds will be assessed for healing and presence of infection.
  Arms: Dressing Removal at 24 Hours
Other: Dressing removal at 48 hours — Dressing will be removed 48 hours after cesarean section and wounds will be assessed for healing and presence of infection.
  Arms: Dressing Removal at 48 Hours

SUMMARY:
The purpose of this study is to assess wound healing at 24 vs 48 hours post cesarean delivery with a modified 1-day ASEPSIS score.

DETAILED DESCRIPTION:
Immediate wound coverage is one of the cornerstones of post-operative wound management. Dressings are typically left in place for 24 to 48 hours following cesarean section to allow ample time for healing and re-epithelialization. The functions of a surgical dressing for wound healing by primary intention are to control postoperative bleeding, absorb exudate, ease pain, and provide protection for newly-formed epithelium. The skin is an important anatomical barrier against microbes; the reformation of an intact epithelial system following injury is an important milestone for the prevention of infection.

Wound healing is a dynamic process that involves the coordinated interaction of a variety of cells, including cytokines, blood cells, extracellular matrix proteins, and parenchyma cells. Wound healing has been artificially divided into three phases: inflammation, tissue formation (proliferation), and tissue remodeling. These phases do not correspond to a precise period of time following injury, and all of the phases overlap to some degree. Re-epithelialization occurs during the proliferation phase and it is defined as the process of restoring an intact epidermis after injury. It involves several processes, including the migration and proliferation of adjacent epidermal keratinocytes into the wound, the differentiation of the neo-epithelium into a stratified epidermis, and the restoration of an intact basement membrane zone (BMZ) that will connect the epidermis and the underlying dermis. Re-epithelialization of wounds begins within hours after injury. Within 24 hours, keratinocytes are actively proliferating from the margins of the wound to cover the defect.

Surgical wounds that are closed by primary intention usually heal rapidly, and re-epithelialization is thought to occur within 24 to 48 hours. Early studies into wound care demonstrated that dressings influence the repair process. The postoperative wound dressing acts to ensure the wound bed stays moist, decrease pain and inflammation, and improve scar appearance. Additionally, occlusive dressings increase the rate of re-epithelialization post-operatively compared to those wounds left open. The importance of dressings has been established, but the ideal time that postoperative dressings should remain in place remains elusive. Studies have shown that early removal of dressings (6 hours after wounding) markedly decreases the rate of resurfacing while leaving the bandage on for greater than 48 hours produced no greater benefit. The United States Centers for Disease Control and Prevention recommends that the sterile dressing stays in place for 24-48 hours postoperatively on an incision that has been closed by primary intention. Although the window of the benefit provided by bandages has not been further refined since these earlier studies. By defining the period during which dressings will promote epithelial resurfacing, our ability to use the dressing optimally will be enhanced.

Our goal of this study is to compared the impact of dressing removal at 24 vs 48 hours on wounds following low-risk cesarean deliveries. While epithelial proliferation begins within hours of closure, it is not at its maximum until 48 to 72 hours following injury. The current standard of care is to keep the dressing in place 24 to 48 hours postoperatively. However, there is no data comparing the optimum timing between 24 and 48 hours. We will, therefore, assess the benefit of leaving the dressing in place for 24 vs 48 hours postoperatively by evaluating its impact on wound appearance and wound score using the ASEPSIS scoring method.

The ASEPSIS is a quantitative scoring method that provides a numerical score related to the severity of wound infection using objective criteria based on wound appearance and the clinical consequences of the infection in 5 days postoperatively. The severity of impaired wound healing is indicated by the total score as follows: satisfactory healing 0 to 10; disturbance of healing 11 to 20; minor wound infection 21 to 30; moderate wound infection 31 to 40; and severe wound infection more than 40. For practical reasons, absolute scores were obtained based on a 1-day reading in our study, rather than the 5-day reading used in the original ASEPSIS scoring system. Another objective of this study is to evaluate patients' satisfaction according to complaints about their incision. Pain, erythema, induration, separation of skin, and serous or purulent exudates will be documented.

ELIGIBILITY:
Inclusion Criteria:

* low-risk obstetric patients aged 18-44 years with term, singleton pregnancies who planned to have Cesarean Delivery (CD).

CD indications:

1. Scheduled nonlabored primary CD for fetal malpresentation,
2. Suspected macrosomia,
3. Maternal request,
4. Placental anomaly,
5. Abnormal / indeterminate fetal heart tracing without labor.
6. First, second, and third repeat CDs will be included.

Exclusion Criteria:

1. Preeclampsia,
2. Preeclampsia with severe features,
3. Eclampsia,
4. Known preoperative infectious disease, any unknown origin preoperative fever,
5. Diabetes,
6. Pregnant with premature rupture of membrane (PROM) or rupture of membrane (ROM),
7. Intraoperative findings suggestive of an underlying cancerous condition,
8. Vertical skin incision,
9. Planned hysterectomy during CD.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 869 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
ASEPSIS Wound Score (1-day) | 24 or 48 Hours Postoperative

SECONDARY OUTCOMES:
ASEPSIS Wound Score (1-day) | 1 Week Follow-Up
ASEPSIS Wound Score (1-day) | 6 Week Follow-Up

OTHER OUTCOMES:
Patients' satisfaction | 24 or 48 Hours Postoperative
Patients' satisfaction | 1 Week Follow-Up
Patients' satisfaction | 6 Week Follow-Up

CONTACTS AND LOCATIONS:
Overall Officials: Gokhan S Kilic, MD, Principal Investigator — The University of Texas Medical Branch, Galveston
Locations (3):
- University of Texas Medical Branch at Galveston, Galveston, Texas, United States
- Turkey (Türkiye) (2):
  - Etlik Zübeyde Hanim Women's Health Training and Research Hospital, Ankara
  - Dicle University, Diyarbakır

REFERENCES:
- [Background] Singer AJ, Clark RA. Cutaneous wound healing. N Engl J Med. 1999 Sep 2;341(10):738-46. doi: 10.1056/NEJM199909023411006. No abstract available. PMID 10471461
- [Background] National Collaborating Centre for Women's and Children's Health (UK). Surgical Site Infection: Prevention and Treatment of Surgical Site Infection. London: RCOG Press; 2008 Oct. Available from http://www.ncbi.nlm.nih.gov/books/NBK53731/ PMID 21698848
- [Background] Li J, Chen J, Kirsner R. Pathophysiology of acute wound healing. Clin Dermatol. 2007 Jan-Feb;25(1):9-18. doi: 10.1016/j.clindermatol.2006.09.007. PMID 17276196
- [Background] Hulten L. Dressings for surgical wounds. Am J Surg. 1994 Jan;167(1A):42S-44S; discussion 44S-45S. doi: 10.1016/0002-9610(94)90010-8. PMID 8109684
- [Background] Eaglstein WH, Davis SC, Mehle AL, Mertz PM. Optimal use of an occlusive dressing to enhance healing. Effect of delayed application and early removal on wound healing. Arch Dermatol. 1988 Mar;124(3):392-5. PMID 3345089
- [Background] HINMAN CD, MAIBACH H. EFFECT OF AIR EXPOSURE AND OCCLUSION ON EXPERIMENTAL HUMAN SKIN WOUNDS. Nature. 1963 Oct 26;200:377-8. doi: 10.1038/200377a0. No abstract available. PMID 14087904
- [Background] Winter GD. Formation of the scab and the rate of epithelisation of superficial wounds in the skin of the young domestic pig. 1962. J Wound Care. 1995 Sep;4(8):366-7; discussion 368-71. No abstract available. PMID 7553187
- [Background] Deodhar AK, Rana RE. Surgical physiology of wound healing: a review. J Postgrad Med. 1997 Apr-Jun;43(2):52-6. PMID 10740722
- [Background] Baum CL, Arpey CJ. Normal cutaneous wound healing: clinical correlation with cellular and molecular events. Dermatol Surg. 2005 Jun;31(6):674-86; discussion 686. doi: 10.1111/j.1524-4725.2005.31612. PMID 15996419
- [Background] Mangram AJ, Horan TC, Pearson ML, Silver LC, Jarvis WR. Guideline for Prevention of Surgical Site Infection, 1999. Centers for Disease Control and Prevention (CDC) Hospital Infection Control Practices Advisory Committee. Am J Infect Control. 1999 Apr;27(2):97-132; quiz 133-4; discussion 96. PMID 10196487
- [Background] Wilson AP, Gibbons C, Reeves BC, Hodgson B, Liu M, Plummer D, Krukowski ZH, Bruce J, Wilson J, Pearson A. Surgical wound infection as a performance indicator: agreement of common definitions of wound infection in 4773 patients. BMJ. 2004 Sep 25;329(7468):720. doi: 10.1136/bmj.38232.646227.DE. Epub 2004 Sep 14. PMID 15367425
- [Background] Wilson AP, Treasure T, Sturridge MF, Gruneberg RN. A scoring method (ASEPSIS) for postoperative wound infections for use in clinical trials of antibiotic prophylaxis. Lancet. 1986 Feb 8;1(8476):311-3. doi: 10.1016/s0140-6736(86)90838-x. PMID 2868173